CLINICAL TRIAL: NCT00282711
Title: The WOMEN Study: What is the Optimal Method for Ischemia Evaluation in WomeN?"A Multi-Center, Prospective, Randomized Study to Establish the Optimal Method for Detection of CAD Risk in Women at an Intermediate-High Pre-Test Likelihood CAD"
Brief Title: The WOMEN Study: What is the Optimal Method for Ischemia Evaluation in WomeN?
Status: Completed | Type: Observational
Sponsor: Hartford Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: HELL001524HE; The WOMEN study
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease; Heart Disease; Coronary Arteriosclerosis; Cardiovascular Disease; Myocardial Ischemia
Keywords: Diagnostic Techniques, Radioisotope; Radionuclide Imaging; Diagnostic Techniques, Cardiovascular; Heart Function tests
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Standard Exercise treadmill test
- 2: Exercise treadmill testing with nuclear imaging

SUMMARY:
The purpose of this study is to compare two types of exercise stress testing to find the best method for detecting heart disease in women.

DETAILED DESCRIPTION:
Coronary artery disease remains the leading cause of morbidity and mortality in women accounting for more than 250,000 deaths per year. While mortality rates have decreased significantly in men during the last several decades, there has been little change for women. Furthermore, despite the high prevalence of ischemic heart disease (IHD) in women, most clinical trials have focused on male cohorts, resulting in a lack of data for women. Their exclusion from clinical trials has been primarily due to the following: 1) child- bearing potential, 2) beyond the arbitrary age limits established for trials, 3) frequent concomitant or advanced disease, and 4) inhomogeneity within the study population.

Extrapolation of the published clinical trial data (predominately obtained in men) for women is controversial due to differences in epidemiology of heart disease in women. Treatment is often sought later in life and is usually accompanied by more advanced disease and co-morbidities, which therefore, impact survival. In addition, women more frequently have an absence of clinical symptoms or an atypical presentation, making the diagnosis of coronary artery disease (CAD) challenging. Furthermore, women may also have their first manifestation of CAD as sudden death or acute myocardial infarction. Therefore, there is a clear need for the early identification of IHD in women so that treatments may be employed prior to having an advanced state of disease and higher risk for unfavorable outcomes.

The optimal non-invasive test for evaluation of IHD in women is unknown. A number of different modalities have been employed including exercise ECG stress testing, 2-dimensional stress echocardiography, single photon emission computerized tomography (SPECT) myocardial perfusion imaging, and electron beam tomography. Additionally, the cohort of women for whom testing is performed is also ill defined.

The most recent AHA/ACC guidelines suggest that ECG stress testing should be the preferred approach. Supportive data for this recommendation are controversial, as many of the studies examining the diagnostic value of ECG stress testing were largely performed in small cohorts of women and are dated. These trials indicate that the diagnostic accuracy of stress testing is only fair (sensitivity=32-89%; specificity=41-68%). A recent meta-analysis in 3,874 women demonstrated modest sensitivity and specificity, 62% and 69% respectively, even after adjustment for referral bias (8). Published guidelines have also included a meta-analysis and confirmed a low level (sensitivity=33%) of detection of disease. Additionally, the high rate of false positives, as well as the inability to fully ascertain the extent of disease, therefore limits the potential value of ECG stress testing.

Even though exercise stress testing is supported by recent clinical guidelines, the addition of SPECT myocardial perfusion imaging has independent and incremental diagnostic and prognostic value. Improved diagnostic accuracy has also been noted with perfusion imaging and its ability to predict cardiac events in women is well established. Furthermore, recent data supports the cost-effectiveness of strategies that employ myocardial perfusion imaging in the assessment of women at risk for ICD.

The current AHA/ACC recommendations fail to take into account that women often have limited ability to complete maximal exercise, a problem that is likely due to their older age and more frequent co-morbidities as compared with men. This functional impairment may lead to a lack of ischemia provocation and/or indeterminate exercise testing results. Maximal predicted heart rate, oxygen consumption, and, more commonly, metabolic equivalents (METs) are measures to estimate physical work capacity. The Duke Activity Status Index (DASI) is a simple 12-item questionnaire that estimates peak oxygen consumption. The Duke Activity Status Index (DASI) questionnaire may identify patients who are likely to perform inadequate exercise, which amounts to nearly 40% of all women referred for exercise testing.

The optimal strategy for the evaluation of women with suspected ischemic heart disease is unknown and quite controversial. Several algorithms have been suggested for the evaluation of women with suspected CAD. A recent consensus paper from the American Society of Nuclear Cardiology suggested a strategy that employed perfusion imaging, but provided little evidence to support such a clinical strategy, such as with a prospective clinical trial. The focus of this investigation is to compare different strategies for the assessment of women at intermediate or high clinical risk for IHD and to do so on a prospective, randomized basis. This study is therefore focused on providing a high level of clinical evidence on which to base future recommendations and guidelines for the care of women with heart disease.

ELIGIBILITY:
Inclusion Criteria:

- Women 60 years of age and older presenting for the evaluation of chest pain, or other anginal equivalent symptoms while at an intermediate-high pretest risk for IHD

Exclusion Criteria:

* Women with known CAD
* Women scoring <5 METs on the DASI
* Nursing or pregnant females
* Nuclear medicine study within the preceding 10 days
* Electrocardiographic abnormalities precluding interpretation of peak stress changes including: Left bundle branch block, electronic ventricular pacemaker, left ventricular hypertrophy, WPW, and resting ST-T wave changes. Additionally, patients currently on digoxin therapy
* Significant valvular heart disease (i.e. severe aortic stenosis or regurgitation, or severe mitral insufficiency)
* Hemodynamic instability (blood pressure >210/110 ml/Hg or <90/60 mm/Hg)
* Left ventricular systolic dysfunction with a left ventricular ejection fraction less than 30 %
* Unavailability for long-term follow-up

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females age 60 and above with suspected heart disease
Sampling Method: Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2004-06; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare 2-year event rates for women capable of performing exercise treadmill testing with normal myocardial perfusion SPECT using Tc-99m tetrofosmin as compared with a negative stress ECG. | 2 years

SECONDARY OUTCOMES:
To evaluate the differential prognostic accuracy of normal exercise myocardial perfusion Tc-99m tetrofosmin SPECT against a normal exercise ECG. | 2 years
To compare the diagnostic sensitivity and specificity of exercise ECG versus exercise ECG-gated Tc-99m tetrofosmin SPECT myocardial perfusion imaging in women who undergo an elective cardiac catheterization. | 2 years
Utility of the DASI questionnaire in determining which women are able to achieve predicted maximal heart rate response with treadmill testing | 2 years
Non-fatal myocardial infarction | 2 years
Unstable angina leading to revascularization | 2 years
Unstable angina with objective evidence of ischemia requiring hospitalization | 2 years
Cardiac death | 2 years
Hospitalization for heart failure | 2 years
Revascularization | 2 years
To provide objective information for developing guidelines for the evaluation of women at intermediate-high likelihood for CAD. | 2 years
A cost-effectiveness analysis will be performed comparing the various evaluation strategies. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary V. Heller, M.D., Ph.D., Principal Investigator — Hartford Hospital, Hartford, CT; Robert C. Hendel, M.D., Principal Investigator — Rush University Medical Center, Chicago, IL; Jennifer H. Mieres, M.D., Principal Investigator — North SHore University Hospital, Long Island, NY; Leslie J. Shaw, Ph.D., Principal Investigator — Atlanta Cardiovascular Research Institute, Atlanta, GA
Locations (42):
- United States (40):
  - Southwest Heart, Tucson, Arizona
  - Cardiology Consultants of Orange Country Medical Group, Inc, Anaheim, California
  - Escondido Cardiology Associates, Escondido, California
  - Mission Internal Medical Group, Mission Viejo, California
  - St. Joseph's Hospital Women's Hrt Cnt, Orange, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sacramento Heart & Vascular Res. Ctr., Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - Cardiovascular Consultants, Walnut Creek, California
  - Hartford Hospital, Hartford, Connecticut
  - Delaware SPECT Imaging, Newark, Delaware
  - Florida Heart Associates, Fort Meyers, Florida
  - Diagnostic Cardiology, PA, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Heart Center, PA, Jacksonville, Florida
  - Jacksonville Heart Center, PA, Jacksonville Beach, Florida
  - Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Cardiac Disease Specialists, Atlanta, Georgia
  - Idaho Cardiology Associates, Boise, Idaho
  - Idaho Cardiology Associates, Meridian, Idaho
  - Fox Valley Cardiovascular Consultants, Aurora, Illinois
  - Saint Francis Hospital of Evanston, Evanston, Illinois
  - Condell Medical Center, Libertyville, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Cardiovascular Associates, Louisville, Kentucky
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Cardiovascular Consultants of Maine, PA, Scarborough, Maine
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Cardiology Associates of Northern Mississippi, Tupelo, Mississippi
  - Cardiovascular Consultants, PC, Kansas City, Missouri
  - Albany Associates in Cardiology, Albany, New York
  - Brooklyn Nuclear SPECT Imaging, Brooklyn, New York
  - Mid-Valley Cardiology, Kingston, New York
  - North Shore University Hospital, Manhasset, New York
  - Blue Stem Cardiology, Bartlesville, Oklahoma
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of SC (MUSC), Charleston, South Carolina
  - Heart Place, Dallas, Texas
  - Deaconess Medical Center, Spokane, Washington
- Canada (2):
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Univ. of Ottawa Heart Insitute, Ottawa, Ontario

REFERENCES:
- [Background] Mieres JH, Shaw LJ, Hendel RC, Miller DD, Bonow RO, Berman DS, Heller GV, Mieres JH, Bairey-Merz CN, Berman DS, Bonow RO, Cacciabaudo JM, Heller GV, Hendel RC, Kiess MC, Miller DD, Polk DM, Shaw LJ, Smanio PE, Walsh MN; Writing Group on Perfusion Imaging in Women. American Society of Nuclear Cardiology consensus statement: Task Force on Women and Coronary Artery Disease--the role of myocardial perfusion imaging in the clinical evaluation of coronary artery disease in women [correction]. J Nucl Cardiol. 2003 Jan-Feb;10(1):95-101. doi: 10.1067/mnc.2003.130362. No abstract available. PMID 12569338
- [Background] Shaw LJ, Miller DD, Romeis JC, Kargl D, Younis LT, Chaitman BR. Gender differences in the noninvasive evaluation and management of patients with suspected coronary artery disease. Ann Intern Med. 1994 Apr 1;120(7):559-66. doi: 10.7326/0003-4819-120-7-199404010-00005. PMID 8116993
- [Background] Mosca L, Grundy SM, Judelson D, King K, Limacher M, Oparil S, Pasternak R, Pearson TA, Redberg RF, Smith SC Jr, Winston M, Zinberg S. Guide to Preventive Cardiology for Women.AHA/ACC Scientific Statement Consensus panel statement. Circulation. 1999 May 11;99(18):2480-4. doi: 10.1161/01.cir.99.18.2480. No abstract available. PMID 10318674
- [Background] Holdright DR, Fox KM. Characterization and identification of women with angina pectoris. Eur Heart J. 1996 Apr;17(4):510-7. doi: 10.1093/oxfordjournals.eurheartj.a014902. No abstract available. PMID 8733082
- [Background] Gibbons RJ, Balady GJ, Beasley JW, Bricker JT, Duvernoy WF, Froelicher VF, Mark DB, Marwick TH, McCallister BD, Thompson PD, Winters WL Jr, Yanowitz FG, Ritchie JL, Cheitlin MD, Eagle KA, Gardner TJ, Garson A Jr, Lewis RP, O'Rourke RA, Ryan TJ. ACC/AHA guidelines for exercise testing: executive summary. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Exercise Testing). Circulation. 1997 Jul 1;96(1):345-54. doi: 10.1161/01.cir.96.1.345. No abstract available. PMID 9236456
- [Background] Hlatky MA, Pryor DB, Harrell FE Jr, Califf RM, Mark DB, Rosati RA. Factors affecting sensitivity and specificity of exercise electrocardiography. Multivariable analysis. Am J Med. 1984 Jul;77(1):64-71. doi: 10.1016/0002-9343(84)90437-6. PMID 6741986
- [Background] Kwok Y, Kim C, Grady D, Segal M, Redberg R. Meta-analysis of exercise testing to detect coronary artery disease in women. Am J Cardiol. 1999 Mar 1;83(5):660-6. doi: 10.1016/s0002-9149(98)00963-1. PMID 10080415
- [Background] Iskandrian AE, Heo J, Nallamothu N. Detection of coronary artery disease in women with use of stress single-photon emission computed tomography myocardial perfusion imaging. J Nucl Cardiol. 1997 Jul-Aug;4(4):329-35. doi: 10.1016/s1071-3581(97)90111-2. No abstract available. PMID 9278880
- [Background] Santana-Boado C, Candell-Riera J, Castell-Conesa J, Aguade-Bruix S, Garcia-Burillo A, Canela T, Gonzalez JM, Cortadellas J, Ortega D, Soler-Soler J. Diagnostic accuracy of technetium-99m-MIBI myocardial SPECT in women and men. J Nucl Med. 1998 May;39(5):751-5. PMID 9591568
- [Background] Hachamovitch R, Berman DS, Kiat H, Bairey CN, Cohen I, Cabico A, Friedman J, Germano G, Van Train KF, Diamond GA. Effective risk stratification using exercise myocardial perfusion SPECT in women: gender-related differences in prognostic nuclear testing. J Am Coll Cardiol. 1996 Jul;28(1):34-44. doi: 10.1016/0735-1097(96)00095-2. PMID 8752792
- [Background] Pancholy SB, Fattah AA, Kamal AM, Ghods M, Heo J, Iskandrian AS. Independent and incremental prognostic value of exercise thallium single-photon emission computed tomographic imaging in women. J Nucl Cardiol. 1995 Mar-Apr;2(2 Pt 1):110-6. doi: 10.1016/s1071-3581(95)80021-2. PMID 9420775
- [Background] Hachamovitch R, Berman DS, Kiat H, Cohen I, Friedman JD, Shaw LJ. Value of stress myocardial perfusion single photon emission computed tomography in patients with normal resting electrocardiograms: an evaluation of incremental prognostic value and cost-effectiveness. Circulation. 2002 Feb 19;105(7):823-9. doi: 10.1161/hc0702.103973. PMID 11854122
- [Background] Galassi AR, Azzarelli S, Tomaselli A, Giosofatto R, Ragusa A, Musumeci S, Tamburino C, Giuffrida G. Incremental prognostic value of technetium-99m-tetrofosmin exercise myocardial perfusion imaging for predicting outcomes in patients with suspected or known coronary artery disease. Am J Cardiol. 2001 Jul 15;88(2):101-6. doi: 10.1016/s0002-9149(01)01601-0. PMID 11448403
- [Background] Shaw LJ, Hendel R, Borges-Neto S, Lauer MS, Alazraki N, Burnette J, Krawczynska E, Cerqueira M, Maddahi J; Myoview Multicenter Registry. Prognostic value of normal exercise and adenosine (99m)Tc-tetrofosmin SPECT imaging: results from the multicenter registry of 4,728 patients. J Nucl Med. 2003 Feb;44(2):134-9. PMID 12571200
- [Background] Marwick TH, Shaw LJ, Lauer MS, Kesler K, Hachamovitch R, Heller GV, Travin MI, Borges-Neto S, Berman DS, Miller DD. The noninvasive prediction of cardiac mortality in men and women with known or suspected coronary artery disease. Economics of Noninvasive Diagnosis (END) Study Group. Am J Med. 1999 Feb;106(2):172-8. doi: 10.1016/s0002-9343(98)00388-x. PMID 10230746
- [Background] Shaw LJ, Heller GV, Travin MI, Lauer M, Marwick T, Hachamovitch R, Berman DS, Miller DD. Cost analysis of diagnostic testing for coronary artery disease in women with stable chest pain. Economics of Noninvasive Diagnosis (END) Study Group. J Nucl Cardiol. 1999 Nov-Dec;6(6):559-69. doi: 10.1016/s1071-3581(99)90091-0. PMID 10608582
- [Background] Gibbons RJ, Chatterjee K, Daley J, Douglas JS, Fihn SD, Gardin JM, Grunwald MA, Levy D, Lytle BW, O'Rourke RA, Schafer WP, Williams SV. ACC/AHA/ACP-ASIM guidelines for the management of patients with chronic stable angina: executive summary and recommendations. A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients with Chronic Stable Angina). Circulation. 1999 Jun 1;99(21):2829-48. doi: 10.1161/01.cir.99.21.2829. No abstract available. PMID 10351980
- [Background] Diamond GA, Forrester JS. Analysis of probability as an aid in the clinical diagnosis of coronary-artery disease. N Engl J Med. 1979 Jun 14;300(24):1350-8. doi: 10.1056/NEJM197906143002402. PMID 440357
- [Background] Chaitman BR, Bourassa MG, Davis K, Rogers WJ, Tyras DH, Berger R, Kennedy JW, Fisher L, Judkins MP, Mock MB, Killip T. Angiographic prevalence of high-risk coronary artery disease in patient subsets (CASS). Circulation. 1981 Aug;64(2):360-7. doi: 10.1161/01.cir.64.2.360. PMID 7249303
- [Background] ACC/AHA 2002 guideline update for exercise testing: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee of Exercise Testing). 2002 American College of Cardiology website. Available at www.acc.org/clinical/guidelines/exercise/dirlndex.htm
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441
- [Derived] Shaw LJ, Mieres JH, Hendel RH, Boden WE, Gulati M, Veledar E, Hachamovitch R, Arrighi JA, Merz CN, Gibbons RJ, Wenger NK, Heller GV; WOMEN Trial Investigators. Comparative effectiveness of exercise electrocardiography with or without myocardial perfusion single photon emission computed tomography in women with suspected coronary artery disease: results from the What Is the Optimal Method for Ischemia Evaluation in Women (WOMEN) trial. Circulation. 2011 Sep 13;124(11):1239-49. doi: 10.1161/CIRCULATIONAHA.111.029660. Epub 2011 Aug 15. PMID 21844080
- See also: ACC/AHA 2002 guideline update for exercise testing: a report of the American College of Cardiology/American Heart Association task Force on Practice Guidelines (Committee of Exercise Testing) — http://www.acc.org/clinical/guidelines/exercise/dirIndex.htm